CLINICAL TRIAL: NCT05066724
Title: Efficacy of Centanafadine SR as a Potential Smoking Cessation Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 405-201-00055
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Centanafadine (Experimental): Participants will receive centanafadine sustained release (SR) tablets, orally at a TDD of 400 milligrams (mg), administered as 200 mg doses, BID, approximately 4 to 6 hours apart, for a total of 7 weeks.
  Interventions: Drug: Centanafadine

INTERVENTIONS:
Drug: Centanafadine — 400 mg total daily dose Centanafadine Sustained Release, oral tablets

SUMMARY:
This study will explore the efficacy and tolerability of centanafadine at a dose of 400 mg per day of centanafadine in promoting smoking abstinence in adult smokers seeking to quit.

DETAILED DESCRIPTION:
This single-group, open-label study of 50 participants will explore the potential of centanafadine in promoting smoking abstinence in adult smokers seeking to quit. The efficacy and tolerability of centanafadine at a dose of 400 mg total daily dose (TDD) (200 mg twice a day (BID)) approximately 4 to 6 hours apart (during a 7-week treatment period) will be compared with a benchmark of abstinence based on historical data from clinical trials of varenicline, viewed as the most efficacious pharmacotherapy currently approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the informed consent form (ICF) and is able to read and understand the information provided in the ICF.
2. Smokers 21 to 65 years of age (inclusive) at screening.
3. Smokes an average of at least 10 commercially available cigarettes per day for the last 12 months.
4. Has an expired air carbon monoxide (CO) reading of at least 10 ppm at screening.
5. At screening, express a desire to quit smoking within the next 30 days.
6. Body mass index (BMI) of 18 to 40 kg/m2, inclusive at screening.
7. Willing and able to comply with the requirements of the study.
8. Owns a smartphone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Participants of childbearing potential (CBP) who are breastfeeding and/or have a positive pregnancy test result.
2. Participant presenting with, or having a history of, uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure > 95 mmHg) or symptomatic hypotension.
3. Participants with known ischemic heart disease or history of myocardial infarction, congestive heart failure (whether controlled or uncontrolled), angioplasty, stenting, coronary artery bypass surgery, or other serious cardiac problems that would place him/her at increased vulnerability to the sympathomimetic effects of stimulant medication.
4. History of seizures (after the age of 17 years).
5. Participants of CBP or sexually active participants unless they agree to practice 2 different methods of birth control or remain abstinent during the course of the trial and for 30 days after the last dose of Investigation Medicinal Product (IMP) for participants of CBP, and 30 days after the last dose of IMP for participants with partners who are of CBP. Unless the participant is sterile (i.e., participants who have had a bilateral oophorectomy or hysterectomy or who have been postmenopausal for at least 12 consecutive months; or participants who have had a bilateral orchidectomy) or remains abstinent, 2 of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pills, birth control injection, birth control implant, birth control patch, condom with spermicide, or sponge with spermicide. Participants who do not agree to refrain from donating sperm from screening through 30 days after the last dose of IMP.
6. Participant has a history of dermatologic adverse reactions secondary to any drug exposure or any active/uncontrolled dermatologic disease.
7. Currently taking antidepressants (e.g., selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs), Tricyclic antidepressants (TCAs), or monoamine oxidase inhibitors (MAOIs)), antipsychotics (such as butyrophenones, thioxanthenes, atypical antipsychotics or other heterocyclics), benzodiazepines, hypnotics, or medications that prolong corrected QT Interval (QTc). MAOI's taken within 30 days of screening.
8. Screening (Visit 1) or Baseline (Visit 2) Columbia-Suicide Severity Rating Scale (C-SSRS) score greater than 0 (any answer "Yes") for the SUICIDAL IDEATION section or greater than 0 for the SUICIDAL BEHAVIOR section (any answer "Yes").
9. Substance use disorder within 12 months prior to screening.
10. Participants that have a positive alcohol test (via breathalyzer or blood), a positive drug screen for illicit drugs (Table 6.3.5) at screening or baseline.

    Participants who test positive for marijuana at screening may be enrolled if they have no evidence of a substance use disorder and if they agree to refrain from use for the duration of the trial.
11. Any participant who has any other medical or physical condition(s) that, in the opinion of the investigator, may prevent the participant from completing the trial or would go against the participant's best interest with participation in the trial. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol.
12. Participants with abnormal laboratory tests, vital sign results, or ECG findings which in the investigator's judgment are medically significant and that would impact the safety of the participant or the interpretation of the trial results.
13. Participants with a history of prior exposure to centanafadine.
14. Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for "Black & Mild" cigars or Cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy, or other smoking cessation treatments (e.g., bupropion as Zyban, or varenicline) within 14 days of screening.
15. Participants who participated in a clinical trial and were exposed to interventional trial medication within the last 30 days prior to screening or who participated in more than 2 interventional clinical trials within the past year.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Rose Research Center
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative centers in the United States from 15 September 2021 to 31 May 2022.
Pre-assignment Details: A total of 287 participants were screened of which 50 participants were enrolled and treated in this study.
Groups:
- Centanafadine: Participants received centanafadine sustained release (SR) tablets, orally, at a total daily dose (TDD) of 400 milligrams (mg), administered as 200 mg doses, twice daily (BID), approximately 4 to 6 hours apart, for a total of 7 weeks.
Period: Overall Study
Arm/Group | Centanafadine
Started | 50
Full Analysis Set (Full Analysis Set included all participants who were administered at least one dose of Investigational Medicinal product (IMP).) | 50
Safety Analysis Set (Safety Analysis Set included all participants who were administered at least one dose of IMP, regardless of any protocol violation.) | 50
Completed | 36
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Non-Compliance With Study Drug | 5
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Enrolled Analysis Set included all participants who signed an informed consent form (ICF) for the trial and were assigned to treatment at the baseline visit.
Groups:
- Centanafadine: Participants received centanafadine SR tablets, orally, at a TDD of 400 mg, administered as 200 mg doses, BID, approximately 4 to 6 hours apart, for a total of 7 weeks.
Arm/Group | Centanafadine
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31
  Black or African American | 12
  Asian | 4
  Other | 1
  Multiple | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Continuous Smoking Abstinence Rate
Description: Participants were considered abstinent from combustible cigarettes if the participant self-reported tobacco abstinence (no cigarette smoking, not even a puff) assessed by responses to daily messages throughout Weeks 4-7. Any participants lost to follow-up after receiving the investigational product, or who have smoked during Weeks 4-7 were counted as non-abstinent. The binomial confidence interval was based on normal approximation. If the number of abstinent or the number of non-abstinent ≤ 5, exact method was used.
Time Frame: Weeks 4 to 7
Population: Full Analysis Set included all participants who were administered at least one dose of IMP.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Centanafadine: Participants received centanafadine SR tables, orally, at a TDD of 400 mg, administered as 200 mg doses, BID, approximately 4 to 6 hours apart, for a total of 7 weeks.
Arm/Group | Centanafadine
Number analyzed (Participants) | 50
percentage of participants | 0 [0.0 to 5.9]

2. Primary Outcome: Percentage of Participants With Continuous Smoking Abstinence Rate Determined Based on Expired Air Carbon Monoxide (CO) Reading Assessed Using the Vitalograph Breath CO Monitor
Description: Participants were considered abstinent from combustible cigarettes if the participants had an exhaled CO level of less than 5 parts per million (ppm) measured using the Vitalograph Breath CO monitor. Participants with actual data that they were smoking (CO value ≥ 5 ppm or any smoking record in self-report) were counted as non-abstinent The binomial confidence interval was based on normal approximation. If the number of abstinent or the number of non-abstinent ≤ 5, exact method was used.
Time Frame: Weeks 4 to 7
Population: Full Analysis Set included all participants who were administered at least one dose of IMP.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Centanafadine
Number analyzed (Participants) | 50
percentage of participants | 2.0 [0.1 to 9.2]

3. Secondary Outcome: Percentage of Participants With Nausea
Description: Nausea was only considered when it was a treatment-emergent adverse event (TEAE). A TEAE is defined as an adverse event (AE) which starts after start of first IMP or an AE continues from baseline of the specific corresponding duration and was serious, trial drug-related or results in death, discontinuation, interruption or reduction of IMP.
Time Frame: From first dose of study drug to 7 days after receiving last dose (Up to Week 8)
Population: Safety Analysis Set included all participants who were administered at least one dose of IMP, regardless of any protocol violation.
Measure: Number; unit: percentage of participants
Arm/Group | Centanafadine
Number analyzed (Participants) | 50
percentage of participants | 12.0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 7 days after receiving last dose (Up to Week 8)
Description: The Safety Analysis Set included all participants who were administered at least one dose of IMP, regardless of any protocol violation.
Arm/Group | Centanafadine
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 35/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Centanafadine (N=50)
Angioedema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Centanafadine (N=50)
Abdominal Pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 5
Mucosal Dryness (General disorders) | 3
Upper Respiratory Tract Infection (Infections and infestations) | 3
Decreased Appetite (Metabolism and nutrition disorders) | 9
Headache (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 11
Drug Eruption (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT05066724/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT05066724/SAP_001.pdf